CLINICAL TRIAL: NCT01786798
Title: Role of Transvaginal Ultrasonography in Evaluating Premenopausal Women Aged More Than 35 Years With Abnormal Uterine Bleeding
Brief Title: Transvaginal Ultrasound in Women With Abnormal Uterine Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RA55/34
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Abnormal Uterine Bleeding
Keywords: Transvaginal sonography; Endometrial thickness; Endometrial pattern; Abnormal uterine bleeding; Endometrial hyperplasia; Endometrial cancer
MeSH Terms: conditions — Metrorrhagia; Endometrial Hyperplasia; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transvaginal sonography (Other)
  Interventions: Device: Transvaginal sonography

INTERVENTIONS:
Device: Transvaginal sonography — Transvaginal sonography will be performed to:
  * measure the endometrial thickness
  * detect the endometrial pattern

SUMMARY:
The objective of this study is to investigate the role of transvaginal ultrasound in detecting endometrial hyperplasia and endometrial cancer in women aged more than 35 presenting with abnormal uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged over than 35
* Abnormal uterine bleeding (menorrhagia/menometrorrhagia/metrorrhagia)
* Accept transvaginal examination (pelvic examination and ultrasound)
* Informed consent

Exclusion Criteria:

* Severe uterine bleeding resulting in unstable vital signs
* Pregnancy
* Current medications: anticoagulants, selective serotonin reuptake inhibitor (SSRI), antipsychotics, corticosteroids, hormones, herbs
* Intrauterine device
* Genital tract pathologies: infection, submucous myoma distorting uterine cavity
* Systemic diseases that may cause coagulopathies: Thyroid disease, liver disease, pituitary/ hypothalamus diseases
* Not able to retrieve endometrial tissue

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy of endometrial thickness and endometrial pattern detected by transvaginal ultrasound in predicting endometrial hyperplasia and endometrial cancer. | 14 months
  The endometrial thickness will be measured in millimeter, at the mid-sagittal plane of the uterus, near the uterine fundus. The measurement will be performed 3 times, from basal layer of the anterior to basal layer of the posterior wall of uterine cavity. The average value of 3 measurements will be used for statistical analysis.
  The endometrial patterns are categorized into 3 groups:
  1. Triple-layer appearance
  2. Mixed echogenic pattern
  3. Hyper-echogenic pattern

SECONDARY OUTCOMES:
To identify the cut-off points of endometrial thickness that can differentiate normal endometrial pathology and endometrial hyperplasia/endometrial cancer. | 14 months
  The results of endometrial thickness will be compared with the endometrial pathologies.The cut-off points of endometrial thickness, in millimeter, that can differentiate normal endometrial pathology and endometrial hyperplasia/endometrial cancer will be analyzed using receiver operating characteristic (ROC) curve.

OTHER OUTCOMES:
To study the prevalence of the various causes of abnormal uterine bleeding in premenopausal women aged more than 35 | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Porntip Sirayapiwat, MD, MSc, Principal Investigator — Department of Obstetrics and Gynecology, Faculty of Medicine, Chulalongkorn University 1873 Rama 4 Road, Patumwan, Bangkok, 10330, Thailand
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Result] Ozdemir S, Celik C, Gezginc K, Kiresi D, Esen H. Evaluation of endometrial thickness with transvaginal ultrasonography and histopathology in premenopausal women with abnormal vaginal bleeding. Arch Gynecol Obstet. 2010 Oct;282(4):395-9. doi: 10.1007/s00404-009-1290-y. Epub 2009 Nov 17. PMID 19921229
- [Result] Getpook C, Wattanakumtornkul S. Endometrial thickness screening in premenopausal women with abnormal uterine bleeding. J Obstet Gynaecol Res. 2006 Dec;32(6):588-92. doi: 10.1111/j.1447-0756.2006.00455.x. PMID 17100821
- [Result] Dueholm M, Jensen ML, Laursen H, Kracht P. Can the endometrial thickness as measured by trans-vaginal sonography be used to exclude polyps or hyperplasia in pre-menopausal patients with abnormal uterine bleeding? Acta Obstet Gynecol Scand. 2001 Jul;80(7):645-51. PMID 11437723